CLINICAL TRIAL: NCT00838396
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Two Period Crossover, Single Dose-Finding Study to Assess the Efficacy and Safety of Controlled Release XP19986 in Patients With Gastroesophageal Reflux Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Controlled Release Arbaclofen Placarbil (XP19986) in Patients With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-B-049
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Eudragit RS; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XP19986 CR (Experimental): On either study Day 1 or study Day 5 (after completion of the minimum 3-day washout period), participants received a single dose of XP19986 10, 20, 40 or 60 mg.
  Interventions: Drug: XP19986 CR
- Placebo for XP19986 CR (Placebo Comparator): On either study Day 1 or study Day 5 (after completion of the minimum 3-day washout period), participants received a single dose of placebo.
  Interventions: Drug: Placebo for XP19986 CR

INTERVENTIONS:
Drug: XP19986 CR
  Other Names: Eudragit RL 100
  Arms: XP19986 CR
Drug: Placebo for XP19986 CR
  Other Names: Sugar Pill
  Arms: Placebo for XP19986 CR

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of arbaclofen placarbil (XP19986) compared to placebo in patients with gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. History of GERD symptoms (e.g. heartburn episodes) at least 3 times per week
2. Discontinuation of drugs used to treat GERD (PPIs, H2-blockers) and/or drugs known to cause GERD symptoms (e.g. nonsteroidal anti-inflammatory drugs [NSAIDs]) for 7 days prior to baseline (Visit 2);
3. Had greater then or equal to 20 postprandial reflux episodes/2 hours recorded using impedance/pH monitoring during Screening/Baseline period (Visit 2)

Exclusion Criteria:

1. History of gastrointestinal disorders other than GERD that may have significantly affected the assessment of reflux episodes or GERD symptoms (e.g. Barrett's Esophagus, active gastric or duodenal ulcer disease, achalasia, scleroderma, etc.).
2. Medical conditions that could have affected assessments of reflux episodes or GERD symptoms (e.g. history of nausea and/or vomiting, neurologic/psychiatric disorders, cardiac disease [e.g. angina], lung disease [e.g. asthma, cough], etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy assessment endpoint of this study was the total number of reflux episodes (acid and non-acid) comparing study drug to placebo | 12 hours

SECONDARY OUTCOMES:
Reflux episodes (acid and non-acid) during each treatment period at various time intervals, dose/exposure to reflux rate relationship, acid reflux events, non-acid reflux events, and GERD symptoms. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jay Huff, M.D., Study Director — XenoPort, Inc.
Locations (3):
- United States (3):
  - Stanford, California
  - Charleston, South Carolina
  - Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No